CLINICAL TRIAL: NCT02486523
Title: Benefits of a Household WASH Package to Community-based Management of Acute Malnutrition (CMAM) Program, Chad
Acronym: OUADINUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Action Contre la Faim (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other); Association Sahélienne de Recherches Appliquées pour le Développement Durable (Other)
Responsible Party: Principal Investigator, Mathias Altmann, Dr, Action Contre la Faim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFI.1836-554994
Record Dates: First submitted 2015-05-26; First posted 2015-07-01 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Severe Malnutrition
Keywords: SAM, severe acute malnutrition
MeSH Terms: conditions — Malnutrition; Severe Acute Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Outpatient management of children diagnosed with severe acute malnutrition.
  Interventions allocated:
  Behavioral: Group discussions after successful discharge Procedure/Surgery: Outpatient Therapeutic Programme
  Interventions: Behavioral: Group discussions after successful discharge; Procedure: Outpatient Therapeutic Programme
- Intervention group (Experimental): Outpatient management of children diagnosed with severe acute malnutrition + "household WASH package"
  Interventions allocated:
  Behavioral: Hygiene promotion sessions Device: Household WASH package The content of the kit: soap and aquatab for 3 months, 20 liters Jerry can, a cup, a plastic kettle for hand washing and the instructions leaflet.
  Behavioral: Household visits during the OTP phase Behavioral: Group discussions after successful discharge Procedure/Surgery: Outpatient Therapeutic Programme
  Interventions: Behavioral: Hygiene promotion sessions; Device: Household WASH package; Behavioral: Household visit; Behavioral: Group discussions after successful discharge; Procedure: Outpatient Therapeutic Programme

INTERVENTIONS:
Behavioral: Hygiene promotion sessions — Hygiene promotion sessions are provided weekly to the caretakers at the health center level. They contain 7 main messages this study is trying to get across: Allocate a protected space for children to play, limiting the likelihood of them ingesting soil or animal feces; Wash the child with soap (hand, face) when outside the protected area; Cleaning and rapid burial of children's stools; Key times for hand washing with soap for the child caretaker; Store drinking water in a closed container located in an elevated place out of reach of animals; Drinking water provided to the child should be treated with chlorine or boiled; Once weaned, avoid giving to the child leftover food, or only after warming it again.
  Arms: Intervention group
Device: Household WASH package — The content of the kit: 200 g soap, aquatab 67 g, 20 liters Jerry can, a cup, a plastic kettle for hand washing and the instructions leaflet.
  Arms: Intervention group
Behavioral: Household visit — A household visit conducted by village's community health volunteers and ACF intervention staff during and after the treatment, to provide refresh training on the messages and the use of the kit.
  Arms: Intervention group
Behavioral: Group discussions after successful discharge — Group discussions on hygiene and care practices with mothers at the community level after successful discharge.
Procedure: Outpatient Therapeutic Programme — Home-based treatment and rehabilitation using Ready-to-use Therapeutic Food (RUTF) for children with severe acute malnutrition

SUMMARY:
The objective of the research is to assess the effectiveness of adding a Household WASH component to the standard outpatient treatment of severe acute malnutrition.

Study design: cluster-randomized controlled trial comparing two interventions:

1. Control group: outpatient management of children diagnosed for severe acute malnutrition only
2. Intervention group: outpatient management of children diagnosed for severe acute malnutrition + "household WASH package"

2000 children, aged between 6 and 59 months, admitted to 20 OTP (Outpatient Therapeutic Program) centers for SAM will be included into the study and followed for 8 months (2 months of treatment, and 6 months after successful discharge).

DETAILED DESCRIPTION:
The Action Contre la Faim (ACF) nutrition project in Kanem started in 2008, and now is set up in 35 health facilities divided across 2 health districts: Mao and Mondo. The management of severe acute malnutrition is done in both OTP (Outpatient Therapeutic Programme) and in TFC (Therapeutic Feeding Center). Between the treatment of SAM in OTPs and TFCs, and the number of curative consultations, the total number of beneficiaries is expected to be 45,065 in 2014 (without double counting).

Clear evidence exists that some Water, Sanitation and Hygiene (WASH) interventions can successfully prevent diarrhea. For instance, interventions aiming at improving water quality at household level or at promoting hand washing with soap do reduce significantly diarrhea incidence. Estimations showed that WASH interventions have a small but measurable benefit on length growth, but not on weight or weight/height. Yet, to our knowledge, no impact of WASH interventions has been assessed, neither during nutritional rehabilitation where children are particularly vulnerable to infections, nor after discharge where immune recovery is still incomplete.

In the context of nutritional rehabilitation of SAM (Severe Acute Malnutrition), the investigators hypothesize that improving water quality and hygiene-related care practices at household level would decrease incidence of WASH-related infections, such as diarrhea, nematode and environmental enteropathy. As such, it would improve weight gain, decrease relapses after successful discharge, and overall, could decrease over time the incidence of acute malnutrition in the community.

The proposed WASH intervention will be added to already existing nutritional activities and it will include: i/ Household water treatment and hygiene kit (water container, water disinfection consumables, soap, cup, hygiene promotion leaflet) provided at beginning of SAM treatment; ii/ sessions of Hygiene promotion provided weekly at health center level iii/ Household visits and hygiene sessions made during the treatment; // group discussion on hygiene and care practices made with mother at community level after successful discharge.

ELIGIBILITY:
Inclusion criteria:

* Children aged between 6 to 59 months
* New admission:

  * Weight for Height Z-score (WHZ) < -3 (WHO2006) or
  * MUAC <115 mm or
  * Presence of bilateral oedema (+ or ++ at OTP admission)
* Other admission:

  * Relapse: after a successful discharge or ≥ 2 months since last visit
  * Re-admission: defaulter < 2 months since last visit
  * Transfer from a stabilization center (SC)
* Caretakers' agreement to participate (through an informed consent)

Exclusion Criteria:

* Signs of medical complications requiring inpatient management,
* Bilateral oedema (+++),
* Transfer from another OTP: treatment already started and child has a identification number (ID) for SAM
* Refusal of caretaker to participate
* Children from families outside the health center coverage

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1572 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Difference in the proportion of post-recovery relapse cases | 2 months and 6 months after successful OTP discharge
  This is a dichotomous variable based on whether a child discharged as cured from the OTP program has a new event of acute malnutrition during the 6 months following the discharge. The relapse proportion for each group = [Total number of relapsing children] / [total number of discharged children that have been followed up] Relative reduction of 42% (from 12% to 7%) is expected.

SECONDARY OUTCOMES:
Difference in the average weight gain at the OTP discharge | an expected average is between 7 and 8 weeks
  The weight gain (g/kg/day) = [weight (g) at discharge - minimum weight (g)] / [Duration from minimum weight to discharge] * [minimum weight (kg)]. The average weight gain (g/kg/day) for each group = [Sum of weight gains of cured children] / [total number of cured children].
  Increase of 3 g/kg/day is expected.
Difference in the anthropocentric measurements (WHZ, HAZ, WAZ) | up to 6 months after OTP discharge
  Weight for Height Z-score (WHZ), Height for age Z-score (HAZ) and Weight for age Z-score (WAZ) and Mid-upper-arm circumference (MUAC) Increase of 0,2 Z-score 6 months after OTP discharge is expected.
Diarrhoea Incidence | up to 6 months follow up
  Loose or watery stools at least three times per day during the week/month prior to the consultation or visit.
Difference in the length of stay in the OTP | an expected average is between 7 and 8 weeks.
  The OTP length of stay is the total number of days spent in the program, from admission of the child to the discharge of a cured child. The average length of stay for all children in each group = [total number of days of cured children] / [number of cured children].
  Reduction of 5 days is expected.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Altmann, Dr, Principal Investigator — ACTION CONTRE LA FAIM | ACF-France
Locations (1):
- Health centers, Mao, Kanem Region, Chad